CLINICAL TRIAL: NCT07398157
Title: Subgaleal Cortical Electrodes in Patients With Parkinson's Disease Undergoing Deep-brain Stimulation Therapy for Sensing and Adaptive Deep-brain Stimulation Over a 24-hour Period.
Brief Title: Simplified, Scalable, 24-hour Adaptive DBS in Parkinson's Disease
Acronym: Subgaleal aDBS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Simon J. Little, MBBS, PhD, Assistant Professor, Clinical Neurology, University of California, San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 25-45027; 1UG3NS140730-01 (NIH)
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: PD - Parkinson's Disease
Keywords: Subgaleal; adaptive; DBS
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinded assessment phase for participants to compare study study-derived adaptive deep brain stimulation to clinically programmed continuous deep brain stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Nighttime adaptive DBS programming (Experimental): The patient will undergo at-home blinded testing of the single power band N2/3 sleep stage aDBS (e.g 75% & 125% conditions, levels chosen for each subject by the clinician or by the study team using data analysis) versus cDBS. Initially the patient will complete ~2 months (60 nights) of randomized, blinded, single night trials of aDBS at lower amplitude (e.g. 75%; 20 nights), aDBS at higher amplitude (e.g. 125% 20 nights) versus cDBS 100% (20 nights) to detect efficacy at the single subject level in independent N-of-1 trials. Stimulation amplitudes will be personalized and selected for tolerability and by searching for amplitudes that impact sleep physiology during the setup phase. Formal final testing will be completed in randomized, counterbalanced condition blocks. Patients will be in cDBS mode during the daytime and will perform a blinded switch to either cDBS or aDBS in the evening before going to sleep (or using the scheduling app).
  Interventions: Device: Medtronic Percept Deep Brain Stimulation (cDBS); Device: Medtronic Percept Deep Brain Stimulation (nighttime aDBS)
- Daytime adaptive DBS Programming (Experimental): We will conduct a blinded, randomized comparison between the effects of aDBS and clinically optimized cDBS on motor signs and symptoms. Both stimulation conditions will be applied for 1 day, in blocks of 2 days that are randomized and counterbalanced for over 40 days in patients' homes. Patients will be in cDBS mode overnight and will perform a blinded switch to either cDBS or aDBS in the morning on waking (these will appear to the patient as programs C and D). We will utilize patients' daily symptom diaries and wearable data. We ask patients to complete the symptom diary (a custom electronic questionnaire) every night before bedtime. The questionnaire focuses on the total number of hours spent with symptoms, symptom severity, and a quality of life (QoL) score validated for daily assessment of health-related QoL (EQ-5D). Evaluated symptoms include the most bothersome and opposite symptom as well as a range of common motor symptoms including bradykinesia, dyskinesia, tremor, etc...
  Interventions: Device: Medtronic Percept Deep Brain Stimulation (cDBS); Device: Medtronic Percept Deep Brain Stimulation (daytime aDBS)
- Open-loop continuous deep brain stimulation (Active Comparator): Participants with Parkinson's disease implanted with Percept and receiving open-loop deep brain stimulation.
  Interventions: Device: Medtronic Percept Deep Brain Stimulation (cDBS); Device: Medtronic Percept Deep Brain Stimulation (daytime aDBS); Device: Medtronic Percept Deep Brain Stimulation (nighttime aDBS)

INTERVENTIONS:
Device: Medtronic Percept Deep Brain Stimulation (cDBS) — Using the Percept pulse generator, patients receive clinically-optimized open loop stimulation to the subthalmaic nucleus.
  Other Names: deep brain stimulation; DBS; cDBS; continuous DBS; continuous deep brain stimulation
Device: Medtronic Percept Deep Brain Stimulation (daytime aDBS) — Using the Percept pulse generator, patients receive daytime adaptive stimulation to the subthalmaic nucleus.
  Other Names: aDBS; adaptive DBS; adaptive deep brain stimulation
  Arms: Daytime adaptive DBS Programming; Open-loop continuous deep brain stimulation
Device: Medtronic Percept Deep Brain Stimulation (nighttime aDBS) — Using the Percept pulse generator, patients receive nighttime adaptive stimulation to the subthalmaic nucleus.
  Other Names: aDBS; adaptive DBS; adaptive deep brain stimulation
  Arms: Nighttime adaptive DBS programming; Open-loop continuous deep brain stimulation

SUMMARY:
The purpose of this study is to test a new way to treat Parkinson's disease (PD). Subjects will be implanted with deep brain stimulator (DBS) devices and electrodes placed under the scalp.

The main questions it aims to answer are:

* Is there a less invasive method to collect useful brain signals? Find out if these brain signals can be related to movement and/or sleep symptoms.
* How to use these brain signals to tailor adaptive deep brain stimulation settings for movement and/or sleep symptoms

Researchers will compare study derived adaptive DBS settings to subject's clinically programmed continuous DBS settings to see which is better at treating patients PD symptoms.

DETAILED DESCRIPTION:
Parkinson's disease (PD) affects 1% of people over 60 years old, is highly disabling and represents a large economic burden. Therapeutic options include dopaminergic replacement and conventional DBS (cDBS) for advanced disease. However, cDBS therapy is currently unresponsive to the dynamic clinical states of patients, resulting in suboptimal control of symptoms during the day. Adaptive DBS (aDBS) seeks to solve this through personalized dynamic modulation of stimulation according to neural signals. Early studies of aDBS (completed by Drs Little, Starr and other research groups) provide proof-of-principle that aDBS can improve motor symptoms and reduce side-effects. Our team has also tested fully embedded, chronic naturalistic aDBS in a randomized, blinded study to show improvements in daytime motor symptoms and quality of life compared to cDBS. Further, we have also recently validated sleep stage specific Non Rapid Eye Movement (NREM) aDBS, that increased cortical slow waves (linked to slowed disease progression). However, full leveraging of these highly promising therapies is currently limited by: 1) Lack of practical (minimally invasive) methods for chronic cortical recordings. 2) Complexity of programming aDBS due to a large parameter space. 3) Fluctuations in neural signals on multiple time scales, including circadian changes and long-term non-stationarity of signals. Our long-term goal is to advance aDBS from specialist research laboratories to real-world clinics through efficient, scalable implementation with the following advances: 1) Reduce risk and complexity of chronic cortical sensing by placing cortical leads in the subgaleal space rather than inside the cranium. 2) Utilize machine learning (ML) and data-driven biomarker and optimization techniques to minimize aDBS programming complexity. 3) Optimize aDBS across the full 24hr cycle - including sleep, with methods for long-term updating of aDBS settings. The study device will be the rechargeable, sensing and aDBS enabled, newly commercially available Medtronic Percept RC DBS system; connected to subgaleal frontal cortex leads and to directional basal ganglia leads. Our UG3 stage will support regulatory approval for Percept RC subgaleal aDBS. In UH3-

1, we will implant 24 PD patients, optimize cDBS, and identify subgroups for daytime and nighttime aDBS. In UH3-2 we will obtain in-clinic and at-home daytime naturalistic neural recordings and perform a blinded evaluation of data-driven chronic aDBS versus cDBS, for treatment of daytime motor fluctuations. In UH3-3, we will obtain in-clinic (sleep lab) and at-home nighttime naturalistic recordings and perform a blinded evaluation of chronic sleep aDBS versus cDBS, to improve NREM sleep duration and increase slow wave amplitude. We anticipate that these techniques will be the basis for a simple "turnkey" aDBS controller, to enable widespread, simple, scaleable and personalized aDBS for the full 24 hr cycle in PD, and provide a rational foundation for adaptive neuromodulation in other neurological and psychiatric diseases.

ELIGIBILITY:
Inclusion criteria

1. Age 25-75.
2. Diagnosis of idiopathic PD.
3. Patient has undergone appropriate therapy with oral medications with inadequate relief as determined by a movement disorders neurologist (Dr. Bledsoe).
4. Patient has requested surgical intervention with deep brain stimulation for their disorder or previous enrollment in sponsored IDE (G220241) to use Percept PC wired to subgaleal sensing, if patients have ongoing daytime fluctuations or sleep dysfunction despite cDBS optimization.
5. Normal preoperative brain MRI.
6. Absence of significant cognitive impairment (score of 24 or greater on the Montreal Cognitive Assessment (MoCA).
7. Signed informed consent.
8. Motor UPDRS-III off medication score 25 to 65 and a >35% improvement with levodopa, predominant rigid/bradykinetic symptoms (ratio of off-medication UPDRS-III limb rigidity/bradykinesia scores to limb tremor scores of >1.2).
9. Motor fluctuations despite optimized medical therapy with at least 2 hours per day of either "off" time, or "on" with dyskinesias.
10. Ability to comply with study follow-up visits for brain recording, testing of closed-loop stimulation, and clinical assessment.

Exclusion criteria

1. Coagulopathy, uncontrolled hypertension, heart disease, or other medical condition considered to place the patient at elevated risk for surgical complications.
2. Patient meets criteria for a psychogenic movement disorder.
3. Pregnancy: all women of childbearing potential will have a negative urine pregnancy test prior to undergoing their surgical procedure.
4. Significant untreated depression (BDI-II score >20) History of suicidal attempt or active suicidal ideation (Yes to #2-5 on C-SSRS).
5. Any personality or mood symptoms that study personnel believe will interfere with study requirements.
6. Patient who requires electroconvulsive therapy, repetitive transcranial magnetic stimulation, or diathermy, implanted neurostimulators and MR-incompatible metallic implants, previous craniotomy on the side of the intended subgaleal implant, and drug or alcohol abuse.
7. Patients who experience adverse effects that are undesirable and detrimental to the health of subjects from DBS or other similar neurostimulators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-11-30 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in number of bothersome movement and/or sleep episodes on adaptive deep brain stimulation compared to open-loop deep brain stimulation | Baseline, aDBS testing, and during Blinded Assessment
  Troublesome movement and/or sleep episodes will be detected using validated home wearable devices along with participant self-reporting.

SECONDARY OUTCOMES:
Change in MDS-UPDRS III scores | Baseline, aDBS testing, and Blinded Assessment
  Change in Movement Disorders Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) III score. The scale consists of 18 items that are each scored 0 to 3, making the total score out of 72 points, with higher scores indicating higher impairment.
Change in Total Electrical Energy Delivered (TEED) | Baseline, aDBS testing, and Blinded Assessment
  Change in TEED calculated using voltage, frequency, pulse width, and impedence values from participant pulse generators, with adaptive compared to open-loop deep brain stimulation (DBS). TEED is measured in microjoules.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Little, Principal Investigator — University of California, San Francisco; Philip Starr, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No